CLINICAL TRIAL: NCT05649319
Title: Effectiveness of Enhanced Recovery After Surgery (ERAS) on Postoperative Recovery After Laparoscopic Distal Gastrectomy: An Open-labeled Randomized Controlled Study
Brief Title: ERAS on Postoperative Recovery After Laparoscopic Distal Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hojin Lee, MD, PhD, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2207-206-1346
Record Dates: First submitted 2022-11-28; First posted 2022-12-14 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Enhanced Recovery After Surgery
Keywords: Enhanced Recovery After Surgery; Stomach Neoplasms; Gastrectomy; Pain, Postoperative
MeSH Terms: conditions — Stomach Neoplasms; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: A prospective randomized open-labeled study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS group (Experimental): Perioperative care for laparoscopic distal gastrectomy is managed according to ERAS protocol.
  Interventions: Procedure: ERAS protocol
- Conventional group (No Intervention): Perioperative care for laparoscopic distal gastrectomy is managed according to our current perioperative practice.

INTERVENTIONS:
Procedure: ERAS protocol — The ERAS protocol involves a pre-admission patient education using audiovisual videos, the reduction of perioperative fasting time with administration of preoperative carbohydrate loading and early resumption of oral feeding after surgery, multimodal postoperative nausea and vomiting prevention, early removal of the nasogastric tube and urinary catheter, and multimodal analgesia to minimize opioid consumption after surgery.
  Arms: ERAS group

SUMMARY:
This prospective, randomized, open-labeled study is designed to evaluate the impact of enhanced recovery after surgery (ERAS) protocol on postoperative quality of recovery in patients undergoing laparoscopic distal gastrectomy. We hypothesize that our ERAS protocol can significantly improve the postoperative quality of recovery in patients with laparoscopic distal gastrectomy.

DETAILED DESCRIPTION:
Adult patients undergoing elective laparoscopic distal gastrectomy are randomly allocated to receive the ERAS protocol (n=49) or conventional protocol (n=49). The conventional groups receive our current perioperative management. The ERAS groups receive our new ERAS protocol including preoperative carbohydrate loading, shortening of perioperative fasting time, and multimodal opioid-sparing analgesia. The primary outcome measure was the postoperative quality of recovery evaluated using the Korean version of Quality of recovery-15 at 24, 48, and 72 hours postoperatively. The secondary outcome measures were pain intensity at rest and during coughing evaluated using an 11-point numeric rating scale at 24, 48, and 72 hours postoperatively, gastrointestinal dysfunction evaluated using the I-FEED score at 24, 48, and 72 hours postoperatively, the occurrence of postoperative nausea and vomiting during the first postoperative 24 hours, postoperative 24 to 48 hour period, and postoperative 48 to 72 hour period, the occurrence of major postoperative complications according to the Clavien-Dindo classification during hospitalization, and length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo elective laparoscopic distal gastrectomy
* American Society of Anesthesiologists (ASA)physical classification I-II
* ECOG Performance Status Scale 0 or 1
* Willingness and ability to sign an informed consent document

Exclusion Criteria:

* Patients with chronic pain
* Gastrectomy with combined resection of other organs
* Patients with history of upper abdominal surgery
* Allergies to anesthetic or analgesic medications (fentanyl, ropivacaine, acetaminophen, NSAIDs)
* Medical or psychological disease that can affect the treatment response

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2023-02-03 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Change of the Quality of recovery-15 during the first 72 hours after surgery | postoperative 24, 48, and 72 hours
  Korean version of Quality of recovery-15 questionnaire (0-150): 0, "very poor recovery"; 150, "excellent recovery"

SECONDARY OUTCOMES:
Postoperative pain score | postoperative 24, 48, and 72 hours
  11-pointed NRS pain score at resting/coughing NRS (0-10): 0,"no pain"; 10, "worst pain imaginable"
Total fentanyl consumption | From the end of surgery to 24, 48, and 72 hours postoperatively
  postoperative fentanyl consumption (mcg) via IV patient controlled analgesia
Postoperative nausea and vomiting | From the end of surgery to 24, 48, and 72 hours postoperatively
  Incidence of postoperative nausea and vomiting (%)
Postoperative gastrointestinal dysfunction | postoperative 24, 48, and 72 hours
  I-FEED score 3 points or more (postoperative gastrointestinal intolerance and dysfunction)
Recovery time | Evaluate every hour starting from 9A on the postoperative day 3 up to discharge
  Postoperative time satisfying the following four criteria: (1) tolerance of soft blended diet (SBD) for 24 h; (2) safe ambulation of 600 m without assistance; (3) Adequate pain control (NRS ≤ 3) with oral non opioid analgesics; and (4) No abnormal physical findings or laboratory test

CONTACTS AND LOCATIONS:
Overall Officials: Do Joong Park, MD, PhD, Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided